CLINICAL TRIAL: NCT04760288
Title: A Phase III, Randomized, Open-Label Study of Pralsetinib Versus Standard of Care for Treatment of RET-Mutated Medullary Thyroid Cancer.
Brief Title: A Study of Pralsetinib Versus Standard of Care (SOC) for Treatment of RET-Mutated Medullary Thyroid Cancer (MTC).
Acronym: AcceleRET-MTC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to several logistical challenges during start-up which could not be overcome study was withdrawn.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO42865; 2020-005269-15 (EudraCT Number)
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Medullary | interventions — pralsetinib; cabozantinib; vandetanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Pralsetinib) (Experimental): Participants will receive pralsetinib at a dose of 400 milligrams (mg) orally once daily (PO QD) in 28-day cycles.
  Interventions: Drug: Pralsetinib
- Arm B (SOC: Cabozantinib/Vandetanib) (Active Comparator): Adult participants will receive investigator's choice of SOC MKI therapy with either 140 mg cabozantinib PO QD or 300 mg vandetanib PO QD in 28-day cycles. Adolescents participants (≥ 12 and < 18 years of age) will receive vandetanib, PO QD or every other day, in 28-day cycles depending on the body surface area (BSA), at a dose determined according to the dosing nomogram available in the E.U. Vandetanib SmPC.
  Interventions: Drug: Cabozantinib; Drug: Vandetanib

INTERVENTIONS:
Drug: Pralsetinib — Participants will receive pralsetinib at a dose of 400 mg, as per the dosing schedule described above.
  Arms: Arm A (Pralsetinib)
Drug: Cabozantinib — Adult participants will receive cabozantinib at a dose of 140 mg, as per the dosing schedule described above.
  Arms: Arm B (SOC: Cabozantinib/Vandetanib)
Drug: Vandetanib — Adult participants will receive vandetanib at a dose of 300 mg and adolescent participants will receive vandetanib as per the dosing schedule described above.
  Arms: Arm B (SOC: Cabozantinib/Vandetanib)

SUMMARY:
A study to evaluate the efficacy and safety of pralsetinib compared with SOC treatment (cabozantinib or vandetanib) for participants with RET (rearranged during transfection)-mutant MTC who have not previously received a SOC MultiKinase Inhibitor (MKI) therapy. Participants will be randomized in a 1:1 ratio into one of two treatment arms: Arm A (pralsetinib) or Arm B (investigator's choice of either cabozantinib or vandetanib for adults and vandetanib for adolescents). Participants whose disease progresses during SOC treatment will be offered the option to cross over to receive pralsetinib after confirmation of progressive disease by blinded independent central review (BICR).

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed unresectable locally advanced or metastatic MTC and be a candidate for systemic therapy with SOC MKI.
* Must have received no prior systemic anticancer treatment with MKI therapies for advanced or metastatic MTC.
* Must have radiologically confirmed progressive disease within the last 14 months and at least one of the following:

  1. A MTC-associated symptom and
  2. CLN (Calcitonin) and CEA (carcinoembryonic antigen) level doubling time of less than 24 months.
* Confirmed RET mutation.
* Must be able to swallow an oral medication.
* Must have an ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use appropriate contraception during the treatment period and for the respective period of time after final dose of study drug.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use appropriate contraception during the treatment period and for the respective period of time after final dose of study drug and to refrain from donating sperm.

Exclusion Criteria:

* Participants who are pregnant or breastfeeding, or intending to become pregnant during the study within 14 days after the final dose of pralsetinib or within 4 months after the final dose of vandetanib or cabozantinib.
* Have disease that is suitable for surgery or radiotherapy administered with curative intent.
* Have been previously treated with any systemic kinase inhibitor therapy regimens, including a selective RET inhibitor, given for recurrent and/or metastatic disease.
* Have received any radiation therapy within 14 days prior to Day 1 of Cycle 1 and any related toxicity must be resolved to Grade 1 or better.
* Participant's tumor has any additional known primary driver alterations other than RET.
* Have known hypersensitivity to pralsetinib, vandetanib, or cabozantinib, or any of their ingredients.
* Have a history of pneumonitis of non-infectious etiology within the last 12 months.
* Have ongoing treatment with chronic immunosuppressants or systemic steroids >10 mg/day.
* Have any history of hereditary bleeding disorder or any evidence of hematemesis.
* Have had major surgery or invasive dental procedure within 3 weeks prior to Day 1 of Cycle 1.
* Have central nervous system (CNS) metastases that are associated with progressive neurologic symptoms, untreated spinal cord compression or requires increasing doses of corticosteroids to control the CNS disease.
* Have clinically significant, uncontrolled, cardiovascular disease.
* Have required treatment with a prohibited medication or herbal remedy.
* Have received hematopoietic growth factor support or transfusion within 14 days of the first dose of study drug.
* Had a major surgical procedure within 14 days of the first dose of study drug.
* Have a history of another primary malignancy that has been diagnosed or required therapy within the past 2 years before randomisation.
* Have a serious infection requiring intravenous (IV) antibiotics within 7 days prior to initiation of study treatment.
* Have an active, uncontrolled infection (viral, bacterial, or fungal) or is positive for Hepatitis B/C infections (HBV/HCV) or HIV.
* Have received organ or allogenic bone marrow or peripheral blood stem cell transplant.
* Is a female who is unwilling to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for at least 4 months after the last dose of study drug.
* Is a male who is unwilling to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for at least 120 days after the final dose of study drug.
* Have prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's or Sponsor's opinion, could affect the safety of the patient or impair the assessment of study results.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2027-10-06 (Estimated); Study Completion 2035-04-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years
  Defined as the time from randomization date to the first documented PD (Progression of Disease), as assessed by BICR according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Time-To-Treatment Failure (TTF) | Up to 13 years
  Defined as the time from randomization date to the discontinuation of study drug during the treatment period due to death, treatment-related adverse event, or PD, as assessed by BICR according to RECIST v1.1, whichever occurs first.
Objective Response Rate (ORR) | Up to 13 years
  Defined as the proportion of participants who achieve a CR (Complete Response) or a PR (Partial Response) prior to progressive disease and/or other anti-cancer therapy, as assessed by BICR according to RECIST v1.1.
Overall Survival (OS) | Up to 13 years
  Defined as the time from randomization date to death due to any cause.
Percentage of Participants With Adverse Events (AEs) | Up to 13 years
  Incidence and severity determined according to the NCI CTCAE v5.0 (National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0) criteria.
Duration of Response (DOR) | Up to 13 years
  Defined as the number of weeks from the time criteria are first met for either a CR or a PR, until the date of documented PD, as assessed by BICR according to RECIST v1.1, or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 13 years
  Defined as the proportion of participants who experience a best response of CR, PR, or stable disease, as assessed by BICR according to RECIST v1.1.
Clinical Benefit Rate (CBR) | Up to 13 years
  Defined as the proportion of participants who experience a CR or a PR or a best response of stable disease with a minimum duration of 6 months, as assessed by BICR according to RECIST v1.1.
Time to Deterioration of Function | Up to 13 years
  Defined as the time from randomization to the date of a participant's first >= 10-point decrease from baseline score, as assessed through the use of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).
Quality of Life (QoL) | Up to 13 years
  Defined as the time from randomization to the date of a participant's first >= 10-point decrease from baseline score, as assessed through the use of the GHS (Global Health Status)/QoL scales.
Acceptability and Palatability of Pralsetinib Capsules | Up to 13 years
  Acceptability Survey scores on Day 1 of Cycle 1 and Crossover Cycle 1 (each cycle is 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).